CLINICAL TRIAL: NCT02860442
Title: Early Intervention to Reduce Alcohol Misuse and Abuse in the Ohio Army National Guard
Brief Title: Project Guard: Reducing Alcohol Misuse/Abuse in the National Guard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keming Gao (Other)
Collaborators: Case Western Reserve University (Other); University of Michigan (Other); University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor-Investigator, Keming Gao, Director, Mood Disorders Program, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 03-16-11; CDMRP-13277015 (Other Grant/Funding Number: U.S. Army Medical Research and Materiel Command)
Record Dates: First submitted 2016-06-07; First posted 2016-08-09 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Use
Keywords: Alcohol misuse; Smartphone app; Screening, Brief Intervention, Referral to Treatment (SBIRT)
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone brief intervention (SP-BI) (Experimental)
  Interventions: Behavioral: Smartphone brief intervention (SP-BI)
- Enhanced Usual Care (EUC) (Placebo Comparator)
  Interventions: Other: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Smartphone brief intervention (SP-BI) — Participants in the SP-BI group will receive a 20-30 minute intervention through an app program based on the FRAMES format: providing personalized Feedback (regarding substance use, risk factors), emphasis on Responsibility for change, Advice, Menu of options, Empathic clinical behaviors, and support of Self-efficacy regarding making changes. The intervention is designed to address the target behavior of alcohol use, and will include a tailored review of participants' goals/values, feedback regarding their alcohol use patterns and consequences (either actual experiences or potential based on risk behaviors), developing a discrepancy between their alcohol use and ability to meet goals and values through a decisional balance exercise, and formulation of a "change plan".
  Arms: Smartphone brief intervention (SP-BI)
Other: Enhanced Usual Care (EUC) — Those assigned to EUC will receive an informational brochure with resources available to members of the military related to mental health and alcohol use. They will be contacted to complete 4-, 8-, and 12-month follow-up assessments.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The overall goal for the study is to test the efficacy of a smartphone app which includes an alcohol brief intervention (SP-BI) versus an Enhanced Usual Care (EUC) condition for National Guard members in the State of Ohio who meet criteria for at-risk drinking in the previous 4 months. The main hypothesis is that those in the SP-BI group with have reduced frequency and intensity of at-risk drinking and fewer binge drinking episodes.

DETAILED DESCRIPTION:
The project is a fully-powered randomized controlled trial of a smartphone app which includes an alcohol brief intervention (SP-BI) versus an Enhanced Usual Care (EUC) condition for National Guard members in the State of Ohio, who are already participating in the Ohio Army National Guard Mental Health Initiative (OHARNG-MHI) study, titled "Resilience and Risk Factors Associated with Deployment Related Posttraumatic Psychopathology", who meet criteria for at-risk drinking in the previous 4 months. After tailoring the content of the SP-BI intervention for NG soldiers, the study will prescreen ~ 8,500 individuals over the three year enrollment period to identify 850participants with at-risk drinking. TParticipants in this study will be randomized to either the SP-BI (n=375) or the EUC condition (n=375) and followed at 4, 8 and 12 months post-enrollment. Participants who are randomized to the SP-BI condition will receive an informational brochure with resources available to members of the military related to mental health and alcohol use and will download a free app on to their smartphones. The app will be developed to be used on both Android and iPhone platforms and will be used over 12 weeks to deliver the study intervention. Those assigned to the EUC condition will receive the informational brochure only.

The specific aims of the study are to compare SP-BI and EUC in: 1) Reducing the frequency and intensity of at-risk drinking at 4 -, 8- and 12-months; 2) Decreasing binge drinking at 4-, 8- and 12 months. The secondary aims are to: 1) Compare the SP-BI and EUC conditions in reducing the frequency of illicit drug use and depressive symptoms at 4-, 8- and 12-months; 2) Examine if deployment status moderates the effect of intervention assignment (SP-BI or EUC) on post-intervention drinking, depressed feelings, and other substance use.

ELIGIBILITY:
Inclusion Criteria:

* Have a past 4-month AUDIT-C score of 5 or more for men and 4 or more for women indicating that they meet criteria for at-risk drinking, AND
* Do not meet any of the exclusion criteria.
* Must be a current or former member of the Ohio Army National Guard (OHARNG) or U.S. Army Reserve based in Ohio.

Exclusion Criteria:

* Those who do not have access to a smart phone with either Android or iOS operating system
* Those in active treatment for substance use disorders (i.e., report addictions treatment in past 4 months) will be excluded because the proposed SBIRT intervention is focused on early brief intervention for those with at-risk drinking and on referral to treatment for those with more serious problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the Number of Drinking Days as Assessed by the Audit-C | Change over time (Baseline, 4-, 8- and 12-months post baseline)
Change in the Number of Drinks per Day as Assessed by the Audit-C | Change over time (Baseline, 4-, 8- and 12-months post baseline)
Change in the Number of Binge Drinking Days as Assessed by the Audit-C | Change over time (Baseline, 4-, 8- and 12-months post baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Blow, PhD, Principal Investigator — Department of Psychiatry, University of Michigan
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT02860442/Prot_SAP_000.pdf